CLINICAL TRIAL: NCT06605040
Title: Audiovisual Materials Disseminated Via Social Media Targeting Evidence-based Rehabilitation Implementation for Physiotherapists
Brief Title: Scientific Content Disseminated Via Social Media for Physiotherapists
Acronym: ASTEROID
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Guilherme Nunes, Adjuct Professor, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4.033.967
Record Dates: First submitted 2024-09-15; First posted 2024-09-20 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Physiotherapy
Keywords: Knowledge translation; continuous education; evidence-based practice

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This protocol outlines a randomized, single-blind (assessors), two-arms, parallel-group controlled trial which will evaluate the the impact of an educational program disseminated via social media compared to plain abstracts send via email on the clinical practice, knowledge and perceptions of physiotherapists. The study outcomes will be categorized into three areas, each of which will be addressed in separate articles: i) effectiveness, including feasibility analysis (quantitative outcomes), ii) qualitative outcomes, and iii) technical outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Social Media (Experimental): The group will receive scientific content via social media
  Interventions: Other: Dissemination via Social Media
- Email (Active Comparator): The group will receive scientific content via email
  Interventions: Other: Dissemination via Email

INTERVENTIONS:
Other: Dissemination via Social Media — Participants in the experimental group will follow a scientific Instagram profile where content will be shared. The profile will remain open, allowing permanent access to all posts. To optimize Instagram's algorithm, we will use an existing active profile. Any control group participants already following the profile will be removed upon allocation.
  For each selected article, we will create three presentations using Instagram features like carousel images and short videos, shared as posts, stories, and reels. This strategy will provide content for 30 weeks of daily posts. Each post will feature visually appealing graphics to convey scientific information and support evidence-based practice (EBP) competencies.
  Arms: Social Media
Other: Dissemination via Email — The participant allocated to the control group will receive a different summary each day, along with a link to the full article. This strategy was chosen to replicate the approach used by scientific journals to disseminate new issues.
  Arms: Email

SUMMARY:
This study is designed to assess how effective social media is in disseminating scientific knowledge to physiotherapists in Brazil. The trial will include physiotherapists who treat at least three patients weekly and regularly use Instagram and WhatsApp. Participants will be randomly assigned to one of two groups: the experimental group will receive scientific content through Instagram, while the control group will receive the same content via email. Both groups will engage with the material for 10 weeks.

The scientific content covers seven key topics related to physiotherapy, such as musculoskeletal and sport rehabilitation, and will be tailored to clinical practice. For the Instagram group, content will be shared via posts, stories, and reels, while the email group will receive summaries and links to full articles. The study aims to evaluate the impact of these interventions on participants' engagement with scientific content and its application to clinical practice.

Key outcomes will include the effectiveness of knowledge dissemination, participant feedback on the audiovisual content, and qualitative insights from interviews. The study will follow a specific timeline, with reassessment three months after the intervention to gauge long-term effects. Data will be analyzed using both quantitative and qualitative methods, ensuring a comprehensive understanding of the intervention's reach and feasibility.

DETAILED DESCRIPTION:
This protocol details a randomized, single-blind controlled trial to assess how effectively scientific content can be disseminated to Brazilian physiotherapists using social media (Instagram). The study will follow physiotherapists who treat at least three patients per week and use Instagram and WhatsApp regularly. These participants will be randomized into two groups: an experimental group receiving content via Instagram and a control group receiving the same information via email.

The study will focus on seven areas relevant to physiotherapy practice, including musculoskeletal rehabilitation, cardiovascular care, and women's health. The content, developed using scientific articles, will be shared daily over 10 weeks. For the Instagram group, the content will be presented through various formats like posts, stories, and reels, with visually engaging elements to boost retention. The email group will receive daily summaries of the articles, similar to a journal-style format.

To maintain participant engagement, both groups will receive weekly summaries, and participants will be assessed on how well they apply the scientific content in practice. The primary outcomes include the effectiveness of content dissemination, participant engagement, and knowledge retention, evaluated through surveys, interviews, and technical assessments. Qualitative interviews will explore participants' experiences, and the quality of the audiovisual materials used will be rated by participants.

The trial will last for 10 weeks, followed by an additional week for reassessment and a three-month follow-up. Data will be analyzed quantitatively to measure the reach and effectiveness of the interventions, with feasibility analyzed using the RE-AIM framework. Qualitative data will be analyzed through thematic analysis, ensuring an in-depth understanding of the intervention's success. This study aims to offer insights into the best methods for delivering scientific knowledge to healthcare professionals via digital platforms.

ELIGIBILITY:
Inclusion Criteria:

* Physiotherapists practicing in Brazil
* Involvement in the rehabilitation of at least three patients per week
* Having access to the social media platforms Instagram and WhatsApp at least once daily on most days of a typical week

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Use of scientific information to make clinical decisions | Baseline and the end of treatment at 10 weeks
  Participants should indicate their level using a scale 0-10 points (0 = I do not use; 10 = I only make clinical decisions using the best available evidence)
Understanding of scientific information interpretation for application in clinical practice | Baseline and the end of treatment at 10 weeks
  Participants should indicate their level using a scale 0-10 points (0 = I do not understand; 10 = I have a complete understanding to apply scientific findings in clinical practice)
Motivation to search for scientific information that could support clinical decisions | Baseline and the end of treatment at 10 weeks
  Participants should indicate their level using a scale 0-10 points (0 = I have no motivation; 10 = I am completely motivated)
Importance of scientific information in making clinical decisions | Baseline and the end of treatment at 10 weeks
  Participants should indicate their level using a scale 0-10 points (0 = No importance; 10 = Extremely important)
Barriers to applying scientific findings | Baseline and the end of treatment at 10 weeks
  Participants will describe their barriers to applying scientific findings in clinical practice and the number of barriers reported will be considered for analysis
Evidence-Based Practice Questionnaire (EBPQ) | Baseline and the end of treatment at 10 weeks
  The EBPQ evaluates EBP competencies and has 24 items scored using a 7-point Likert scale (1-7 points); mean of the items will be used for analysis
Overcoming the reported barriers | End of treatment at 10 weeks
  Participants will be asked whether the program helped to overcome the reported barriers (yes or no answer)

OTHER OUTCOMES:
Completion | End of treatment at 10 weeks
  Number of participants who completed the study
Level of participation | End of treatment at 10 weeks
  Participants should indicate their level using a scale 0-10 points (0 = I did not pay attention to any shared material; 10 = I read all the shared material of my interest)
Impact of program on the clinical practice and decisions | End of treatment at 10 weeks
  Participants should indicate their level using a 5-point Likert scale (1=much worse, 2= worse, 3=the same, 4= better, 5=much better)
Use of shared information | End of treatment at 10 weeks
  Participants will indicate whether they applied information shared during the program in clinical practice (yes or no answer)
Influence of the program | End of treatment at 10 weeks
  Participants will indicate whether the program Influenced them to do something different in clinical practice (yes or no answer)
Intervention's modification | During the whole program which will take approximately 7 months
  We will register whether modifications to the interventions are necessary during the study
Contamination of control group | During the 10 weeks of treatment
  Checking if participant is following the Instagram's profile
Attitude towards seeking information from channels that facilitate the understanding of high-quality scientific findings | End of treatment at 10 weeks
  Participants should indicate their level using a scale 0-10 points (0 = I will not use such information source; 10 = I will definitely use information source that facilitate my understanding)
Approach to study | End of treatment at 10 weeks
  Participants will indicate whether the program influenced on the approach to studying technical content (yes or no answer)
Use of channels to facilitate understanding | 3-month follow-up
  Participants will indicate whether they have used channels that facilitate the understanding of scientific findings
Application of information from different channels | 3-month follow-up
  Participants will indicate whether they have applied information from channels that facilitate the understanding of scientific findings in clinical practice
Qualitative outcome | End of treatment at 10 weeks
  Semi-structured interviews aimed at understanding their perceptions of the application of scientific content in clinical practice and their views on the interventions. Individual interviews will be conducted via telephone or video call, with responses to open-ended questions being audio-recorded.
Quality of information | End of treatment at 10 weeks
  Participants should indicate their opinion about the quality of information using a scale 0-10 points (0 = terrible content; 10 = excellent content)
Visual quality of the shared materials | End of treatment at 10 weeks
  Participants should indicate their opinion using a scale 0-10 points (0 = worst visual quality; 10 = excellent visual quality)
Metrics from social media | During the whole program which will take approximately 7 months
  We will collect engagement metrics from Instagram

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme S Nunes, PhD, Principal Investigator — Universidade Federal de Santa Maria
Locations (1):
- Federal University of Santa Maria, Santa Maria, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No